CLINICAL TRIAL: NCT01887886
Title: A Randomized, Phase III, Multicenter, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of Onartuzumab in Combination With Erlotinib as First-Line Treatment for Patients With MET-Positive Unresectable Stage IIIb or IV Non-Small Cell Lung Cancer (NSCLC) Carrying an Activating EGFR Mutation
Brief Title: A Study of Onartuzumab in Combination With Erlotinib in Patients With MET-Positive Stage IIIB or IV Non-Small Cell Lung Cancer Carrying an Activating Epidermal Growth Factor Receptor (EGFR) Mutation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GO28758; 2013-000868-29 (EudraCT Number)
Record Dates: First submitted 2013-06-25; First posted 2013-06-27 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — Erlotinib Hydrochloride; onartuzumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Onartuzumab + Erlotinib (Experimental)
  Interventions: Drug: erlotinib; Drug: onartuzumab
- Placebo + Erlotinib (Active Comparator)
  Interventions: Drug: erlotinib; Drug: placebo

INTERVENTIONS:
Drug: erlotinib — 150 mg orally daily
Drug: onartuzumab — 15 mg/kg IV every 3 weeks
  Arms: Onartuzumab + Erlotinib
Drug: placebo — IV every 3 weeks
  Arms: Placebo + Erlotinib

SUMMARY:
This multicenter, randomized, double-blind, placebo-controlled study will evaluate the safety and efficacy of onartuzumab in combination with erlotinib in patients with previously untreated, unresectable stage IIIB or IV non-small cell lung cancer identified to carry and activating EGFR mutation and MET-positive. Patients will be randomized to receive either onartuzumab 15 mg/kg intravenously every 3 weeks in combination with erlotinib 150 mg orally daily or placebo in combination with erlotinib. Anticipated time on study treatment is until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, >/= 18 years of age
* Histologically confirmed, unresectable Stage IIIB or IV non-small cell lung cancer (NSCLC)
* No prior treatment for unresectable Stage IIIB or IV NSCLC
* Measurable radiographic evidence of disease according to RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Prior exposure to agents targeting either the Hepatocyte Growth Factor (HGF) or MET pathway
* Exposure to an investigational or marketed agent that can act by EGFR inhibition
* Pleural effusion, pericardial fluid, or ascites requiring drainage every other week or more frequently
* Brain metastasis or spinal cord compression not definitively treated with surgery and/or radiation, or previously diagnosed and treated central nervous system (CNS) metastases or spinal cord compression without evidence of clinically stable disease for >/=4 days. Note: Patients with treated CNS metastases who are asymptomatic and on a stable dose of corticosteroids for >/= 14 days prior to randomization are eligible.
* History of another malignancy in the previous 5 years, unless cured by surgery alone and continuously disease-free
* Radiographically evident interstitial lung disease , concurrent infection, or a history of any of these conditions
* Inadequate hematologic, biochemical, and organ function
* Pregnant or lactating women
* Life expectancy of < 12 weeks
* Receipt of an investigational drug within 28 days prior to initiation of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (investigator-assessed according to RECIST v1.1) | approximately 3 years

SECONDARY OUTCOMES:
Overall survival | approximately 3 years
Overall response rate | approximately 3 years
Time to deterioration (>/= 10 points [transformed score] from baseline) in patient-reported lung cancer symptoms | approximately 3 years
Patient reported outcomes: HRQoL/EORTC QLC-C30/EORTC QLQ-LC31 questionnaires | approximately 3 years
Safety: Incidence of adverse events | approximately 3 years
Pharmacokinetics: Area under the concentration-time curve (AUC) | Day 1 Cycles 1, 2 and 4

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (30):
- United States (14):
  - Bakersfield, California
  - Fullerton, California
  - Long Beach, California
  - Los Angeles, California
  - San Luis Obispo, California
  - Fort Myers, Florida
  - Orlando, Florida
  - St. Petersburg, Florida
  - Chicago, Illinois
  - Marrero, Louisiana
  - Metairie, Louisiana
  - St Louis, Missouri
  - Canton, Ohio
  - Nashville, Tennessee
- France (3):
  - Caen
  - Lyon
  - Nantes
- Germany (3):
  - Großhansdorf
  - Oldenburg
  - Villingen-Schwenningen
- Japan (3):
  - Ehime
  - Okayama
  - Yamaguchi
- Tanjung Bungah, Malaysia
- South Korea (2):
  - Gwangju
  - Suwon
- Spain (2):
  - Barcelona, Barcelona
  - Madrid, Madrid
- Taiwan (2):
  - Taichung
  - Taipei